CLINICAL TRIAL: NCT00148148
Title: Phase II Randomised Study of the Safety, Efficacy and Pharmacokinetics of Caspofungin (CAS), Liposomal Amphotericin B (LAMB) or the Combination of Caspofungin With Liposomal Amphotericin B for Patients After Stem-Cell Transplantation
Brief Title: A Study of Caspofungin, Liposomal Amphotericin B or the Combination of Both for Patients After Stem-Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKS-MS-005-KMT-10/03; BfArM 4021825
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2007-01

CONDITIONS: Hematopoietic Stem Cell Transplantation; Fungus Diseases
Keywords: Hematopoietic Stem Cell Transplantation; Caspofungin; Liposomal Amphotericin B
MeSH Terms: conditions — Mycoses | interventions — Caspofungin; liposomal amphotericin B

INTERVENTIONS:
Drug: caspofungin
Drug: liposomal amphotericin B

SUMMARY:
The study compares the safety, efficacy and pharmacokinetics of caspofungin, liposomal amphotericin B or the combination of both in the antifungal treatment of adult patients after allogeneic haematopoietic stem-cell transplantation with granulocytopenia and persistent i.g. recurrent fever under adequate antibacterial therapy.

DETAILED DESCRIPTION:
This is an open, randomised, three-arm multicenter phase II clinical trial investigating the safety, tolerance and plasma pharmacokinetics of caspofungin, liposomal amphotericin B and the combination of both agents as empirical antifungal therapy in adult patients following allogeneic hematopoietic stem cell transplantation.

Eligible patients are those with profound granulocytopenia (≤ 500 neutrophil granulocytes) and persistent or recurrent fever despite broad-spectrum antibacterial therapy of a minimum of 36-48 hours duration. Patients are stratified according to the type of the transplantation (human leukocyte antigen [HLA] matched/related versus HLA-mismatched/unrelated) and randomized into one of the following treatment arms: Caspofungin alone (50 mg/day with a loading dose of 70 mg on day 1), liposomal amphotericin B alone (3 mg/kg/day), or the combination of caspofungin and liposomal amphotericin B (similar dosages as in the single-drug treatment arms).

Caspofungin and liposomal amphotericin B are administered once daily as an intravenous infusion. Serial plasma samples for determination of pharmacokinetic parameters are collected on days one and four of treatment. Safety and tolerance of the randomised intervention are evaluated daily, following the last dose of study drug and at 14 days after last dose of study drug according to current NCI-CTC criteria. Antifungal efficacy and survival are evaluated following the last dose of study drug and at 14 days after the last dose of study drug.

Treatment with study drug is continued until either:

1. treatment limiting intolerance or toxicity;
2. hematopoietic engraftment (≥ 500 neutrophil granulocytes on three consecutive days) and defervescence; or
3. the occurrence of a probable or proven invasive fungal infection using current EORTC/MSG criteria.

Febrile granulocytopenic patients with probable or proven invasive fungal infections are not eligible for this study. Patients who develop a probable or proven breakthrough infection are taken off study and receive standard therapy. Breakthrough infections are defined as probable or proven invasive fungal infections that occur during treatment with study medication.

Twenty-five patients with a minimum duration of treatment of four days will be randomised per study arm. Patients who receive at least one dose of study drug are eligible for analysis of safety, tolerance and pharmacokinetics. For the analysis of the secondary endpoints of antifungal efficacy and survival, two separate cohorts will be analysed. These include:

1. patients who received at least one dose of study drug; and
2. patients who received ≥ four doses of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> or = 18 years of age) with granulocytopenia (absolute number of neutrophil granulocytes [ANC]: < or = 500/µL) who have undergone allogeneic haematopoeitic stem cell transplantation and immunosuppression with cyclosporin A
* Patients with persistent or recurrent fever (oral temperature > or = 38.0°C) and granulocytopenia (absolute neutrophil count < or = 500/µL) and adequate antibacterial therapy for > or = 36-48 hours, who need empirical antimycotic therapy
* Already inserted at least double-lumen central venous catheter for administration of drugs and extraction of plasma samples
* Sufficient renal and hepatic function
* Availability of negative pregnancy test and adequate contraceptive measures for female patients of childbearing age
* Availability of written informed consent from the patient or respectively from the legal representative after prior information

Exclusion Criteria:

* Patients with active, possible or proven (MSG-EORTC criteria) invasive fungal infection at time of enrollment
* Pregnant or nursing patients
* Patients with pathological functional renal or hepatic parameters
* Patients with clinical or laboratory chemical evidence of active veno-occlusive disease (VOD)
* Hemodynamically unstable patients with a life expectancy of less than 5 days
* Patients undergoing co-medication with rifampicin, phenytoin, carbamazepine, phenobarbital, dexamethasone, efavirenz and nevirapine
* Patients with prior known serious reaction to echinocandin-antifungal formulation or documented allergy to amphotericin B
* Patients with other condition or illness which, in the estimation of the investigator, distorts the study results or leads to an additional risk for the patient
* Prior inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2004-05; Study Completion 2007-12

PRIMARY OUTCOMES:
Safety and efficacy of caspofungin, liposomal amphotericin B and the combination of caspofungin with liposomal amphotericin B in accordance with NCI-CTC toxicity

SECONDARY OUTCOMES:
Pharmacokinetics and recording of the dose-intensity of caspofungin and liposomal amphotericin B in the setting of allogeneic stem cell transplantation
Examination of pharmacokinetical interactions between caspofungin and liposomal amphotericin B
Recording of the efficacy of caspofungin, liposomal amphotericin B and the combination of caspofungin and liposomal amphotericin B in the case of empirical antimycotic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Groll, M.D., Principal Investigator — University Hospital Muenster
Locations (1):
- KKS Münster University Hospital, Münster, North Rhine-Westphalia, Germany